CLINICAL TRIAL: NCT01604655
Title: ProspEctive Randomized First Evaluation in Chest Pain Trial
Brief Title: ProspEctive First Evaluation in Chest Pain Trial
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-307
Record Dates: First submitted 2012-05-17; First posted 2012-05-24 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Chest Pain; Shortness of Breath; Suspected Acute Coronary Syndrome
Keywords: Chest pain; shortness of breath; suspected acute coronary syndrome; stress testing; coronary computed tomography angiography
MeSH Terms: conditions — Chest Pain; Dyspnea | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronary CT Angiography (Active Comparator): Patient admitted with chest pain is randomized to CCTA for assessment.
  Interventions: Procedure: Coronary CT Angiography
- Stress Test (Active Comparator): Patients admitted with chest pain are randomized to a stress test (stress SPECT or Echocardiography) for assessment.
  Interventions: Procedure: Stress Test

INTERVENTIONS:
Procedure: Coronary CT Angiography — CCTA
  Arms: Coronary CT Angiography
Procedure: Stress Test — Stress Test
  Arms: Stress Test

SUMMARY:
The purpose of this study is to determine the best initial test in patients admitted to the hospital complaining of chest pain.

DETAILED DESCRIPTION:
Currently, physicians can either choose a stress test or a CT scan of the heart to evaluate patients admitted with with chest pain. Very little is known about which test provides the best information to physicians, positively impacts patients medical care, and decreases future hospital admissions and testing. To study this the investigators are randomizing patients admitted to our hospital with chest pain to a stress test or coronary CT angiography. The investigators will then follow these patients for a 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain or SOB admitted for rule out acute coronary syndrome
* Age ≥45 years
* EKG non-diagnostic for acute coronary syndrome
* At least 1 set of negative troponin I

Exclusion Criteria:

* Patient with ST elevation myocardial infarction.
* Patients with non-ST elevation myocardial infarction.
* Patients with known CAD.
* Patients with serum creatinine > 1.5.
* Atrial fibrillation or marked irregular heart rhythm.
* Patients in whom heart rate cannot be controlled.
* Patient with allergies to iodinated contrast agents.
* Pregnant women
* Patients unable to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to discharge | Initial hospitalization
Change in medical regimen | Initial hospitalization
Downstream cardiovascular testing and hospitalization | 2 years

SECONDARY OUTCOMES:
All-cause mortality | 7 days, 30 days, 6, 12, and 24 months.
  This measure is to ascertain if CCTA and stress testing can be used safely as the initial test in patients admitted to the hospital with chest pain.
Cardiovascular mortality | 7 days, 30 days, 6, 12, and 24 months.
  This measure is to ascertain if CCTA and stress testing can be used safely as the initial test in patients admitted to the hospital with chest pain.
Non-fatal myocardial infarction | 7 days, 30 days, 6, 12, and 24 months.
  This measure is to ascertain if CCTA and stress testing can be used safely as the initial test in patients admitted to the hospital with chest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Uretsky, MD, Principal Investigator — St. Luke's and Roosevelt Hospital Centers
Locations (1):
- St. Luke's and Roosevelt Hospitals, New York, New York, United States

REFERENCES:
- [Derived] Uretsky S, Argulian E, Supariwala A, Agarwal SK, El-Hayek G, Chavez P, Awan H, Jagarlamudi A, Puppala SP, Cohen R, Rozanski A. Comparative effectiveness of coronary CT angiography vs stress cardiac imaging in patients following hospital admission for chest pain work-up: The Prospective First Evaluation in Chest Pain (PERFECT) Trial. J Nucl Cardiol. 2017 Aug;24(4):1267-1278. doi: 10.1007/s12350-015-0354-6. Epub 2016 Apr 5. PMID 27048306